CLINICAL TRIAL: NCT02716506
Title: Finnish Pelvic Organ Prolapse Surgery Survey 2015: Incidence, Methods, Complications and Effect on Quality of Life of Pelvic Organ Prolapse Operations in Finland in 2015
Brief Title: FINPOP 2015: Incidence, Methods, Complications and Quality of Life of Pelvic Organ Prolapse Operations in Finland 2015
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Society for Gynecological Surgery in Finland (Other)
Responsible Party: Principal Investigator, Nina Mattsson, MD, Society for Gynecological Surgery in Finland
Other Study IDs: Finpop 2015
Record Dates: First submitted 2015-11-10; First posted 2016-03-23 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: POP surgery
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic POP: POP surgery in year 2015
  Interventions: Procedure: POP surgery

INTERVENTIONS:
Procedure: POP surgery — Any surgical procedure that is done to treat the symptomatic POP

SUMMARY:
The aim of this study is to investigate the safety and effectivity of pelvic organ prolapse (POP) surgery. In this multi center study the population consists of POP operations done in Finland year 2015.The study is prospective and validated questionnaires are used to measure the symptoms of POP and the quality of life before and six months after the operation. Methods and complications of surgery are reported by doctors in all 40 participant hospitals.

DETAILED DESCRIPTION:
Patients awaiting for surgical procedure for a symptomatic pelvic organ prolapse (POP) are recruited for the study. The recruiting is done in 41 hospitals in Finland, at gynecological outpatient clinics. Participants are given information of the study and give a written approval to join the study. Participants are asked to fill in questionnaires, that measure the quality of life. Three validated questionnaires are used: Pelvic Floor Distress Inventory PFDI-20, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire PISQ-12 and health-related quality of life instrument 15D. These questionnaires are sent to participants 6 months, 2 and 5 years after the surgical treatment. The participants are also asked to report adverse effects related to the treatment and their satisfaction to the treatment. Information about the surgical procedure (i.e. type and duration of the procedure, blood loss, antibiotic and thrombosis prophylaxis) by the operating doctors. Both immediate and delayed treatment-related adverse effects are also reported by the doctors. Data is partly collected by questionnaires filled in internet. All the collected data is protected by high security and coded before analyses. Permission of protocol used in this study is given by the Ethical Committee of University of Eastern Finland and Finnish National Institute for Health and Welfare.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pelvic organ prolapse
* Mental and psychological ability to understand the study information and to give an approval
* Knowledge of Finnish or Swedish language

Exclusion Criteria:

* Other than Finnish or Swedish language
* Psychological disability to understand the study information

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a symptomatic pelvic organ prolapse (POP) operated in year 2015 in Finland
Sampling Method: Probability Sample
Enrollment: 3515 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2025-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Härkki, PhD, Study Chair — Finnish Society of Gynecological Surgery
Locations (1):
- UEF, Kuopio, Eastern Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wihersaari O, Karjalainen P, Tolppanen AM, Mattsson N, Jalkanen J, Nieminen K. Prolapse recurrence, methods of reoperation, and long-term mesh complications-A nationwide follow-up study. Acta Obstet Gynecol Scand. 2025 Nov 24. doi: 10.1111/aogs.70083. Online ahead of print. PMID 41277806
- [Derived] Wihersaari OAE, Karjalainen P, Tolppanen AM, Mattsson N, Nieminen K, Jalkanen J. Quality of Sexual Life Before and After Pelvic Organ Prolapse Surgery. Urogynecology (Phila). 2024 Oct 1;30(10):838-846. doi: 10.1097/SPV.0000000000001568. PMID 39752612

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic POP
Started | 3515
6 Months | 2528 (Patients that completed the questionnaires six months after the operation.)
2 Years | 2351 (Patients that completed the questionnaires two years after the operation.)
Completed | 2351
Not Completed | 1164

BASELINE CHARACTERISTICS:
Groups:
- Symptomatic POP: Patients that were operated for POP in 2015 in Finland and participated the study
Arm/Group | Symptomatic POP
Number analyzed (Participants) | 3512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1764
  >=65 years | 1748
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3512
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 3512

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life After the POP Surgery
Description: Quality of life is measured by using 15 dimensional quality of health measurement instrument. Minimum value is 0 and maximum value is 1. Higher scores mean better outcome.
Time Frame: 24 months after the surgery
Population: Analysis of the patients who answered the 15-D questionnaire 24 months after the operation.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Symptomatic POP
Number analyzed (Participants) | 2314
units on a scale | 0.898 [0.894 to 0.902]

2. Secondary Outcome: Symptoms Related to Pelvic Organ Prolapse
Description: Condition-specific questionnaire Pelvic Floor Distress Inventory (PFDI-20) is used. Minimum value is 0 and maximum value is 300. Higher scores mean more bothersome symptoms.
Time Frame: 24 months after the surgery
Population: Change in PFDI-20 scores 24 months after the operation compared to the baseline scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic POP
Number analyzed (Participants) | 2342
score on a scale | 49.24 (44.61)

ADVERSE EVENTS:
Arm/Group | Symptomatic POP
All-Cause Mortality (participants affected / at risk) | 0/3512
Serious Adverse Events (participants affected / at risk) | 15/3512
Other Adverse Events (participants affected / at risk) | 353/3512
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symptomatic POP (N=3512)
Serious adverse event (Clavidien dindo IV) (Surgical and medical procedures) | 15 (15) — Clavidien dindo classification
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symptomatic POP (N=3512)
Minor adverse events (Surgical and medical procedures) | 353 (353) — Clavidien dindo I-III

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No